CLINICAL TRIAL: NCT06763094
Title: Efficacy of Calcium Dobesilate As an Alternative Method for Treatment of Menorrhagia, Comparison to Tranexamic Acid
Brief Title: Efficacy of Calcium Dobesilate Versus Tranexamic Acid for Treating Heavy Menstrual Bleeding
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Bazgha Naeem, Post Graduate Resident, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exp127
Record Dates: First submitted 2024-12-21; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Menorrhagia; Abnormal Uterine Bleeding
MeSH Terms: conditions — Menorrhagia; Metrorrhagia | interventions — Calcium Dobesilate; Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Patients receiving Calcium Dobesilate (Doxium) (Active Comparator): Intervention: Patients in Group A will be administered Calcium Dobesilate (Doxium) capsules.
  Dosage: The dose will be 500 mg of Calcium Dobesilate, administered orally at a frequency of three times a day. The total daily dose can range from 1-4 tablets (equivalent to 0.5-2 g/day), starting from the first day of the menstrual cycle and continuing until the bleeding ceases.
  Interventions: Drug: Calcium dobesilate (Doxium)
- Group B: Patients receiving Tranexamic Acid (Active Comparator): Intervention: Patients in Group B will receive Tranexamic Acid capsules. Dosage: The dose will be 500 mg of Tranexamic Acid, administered orally at a frequency of three times a day. This will continue from the first day of the menstrual cycle until the bleeding stops.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Calcium dobesilate (Doxium) — This intervention is unique because Calcium Dobesilate is not a hormonal agent and does not carry the risks associated with hormonal therapies, such as potential impact on fertility or long-term endocrine effects. Additionally, it may be more suitable for patients who cannot tolerate hormonal treatments due to contraindications such as previous thrombotic events or risk factors for thrombosis.
  Arms: Group A: Patients receiving Calcium Dobesilate (Doxium)
Drug: Tranexamic Acid — Tranexamic Acid stands out due to its non-hormonal action in managing menorrhagia, providing an alternative for women who are contraindicated for hormonal treatments or prefer non-hormonal solutions. Unlike other hormonal treatments, Tranexamic Acid does not impact fertility or have significant endocrine effects.
  Arms: Group B: Patients receiving Tranexamic Acid

SUMMARY:
The goal of this clinical trial is to determine if calcium dobesilate is an effective alternative to tranexamic acid for treating menorrhagia in women aged 18 to 39 years. The main questions it aims to answer are:

Does calcium dobesilate reduce menstrual blood loss and improve hemoglobin levels as effectively as tranexamic acid? What side effects and acceptability differences exist between calcium dobesilate and tranexamic acid? Researchers will compare calcium dobesilate to tranexamic acid to see if calcium dobesilate is as effective in reducing heavy menstrual bleeding and improving patient outcomes.

Participants will:

Take calcium dobesilate or tranexamic acid during their menstrual cycle for three consecutive cycles.

Record menstrual blood loss using the Pictorial Blood Loss Assessment Chart (PBAC).

Attend follow-up visits after each menstrual cycle to monitor hemoglobin levels, menstrual symptoms, and any side effects.

DETAILED DESCRIPTION:
This randomized controlled trial aims to compare the efficacy and safety of calcium dobesilate and tranexamic acid in treating menorrhagia in women aged 18 to 39 years. Menorrhagia, characterized by heavy menstrual bleeding exceeding 80 mL per cycle, significantly impacts quality of life and may lead to complications such as anemia.

Participants meeting the inclusion criteria will be randomly assigned to one of two groups:

Group A: Participants will receive calcium dobesilate (500 mg capsules), administered orally at a daily dose of 0.5-2 g during each menstrual cycle for three consecutive cycles.

Group B: Participants will receive tranexamic acid (500 mg capsules), administered orally at a dose of two capsules three times daily during each menstrual cycle for three consecutive cycles.

Primary outcomes will include:

Reduction in menstrual blood loss as measured by the Pictorial Blood Loss Assessment Chart (PBAC).

Improvement in hemoglobin levels after three cycles. Arrest of bleeding after discontinuation of the medications. Secondary outcomes will focus on the acceptability of treatment and side effects, such as nausea, headache, and gastrointestinal discomfort.

Data will be collected through patient records, physical examinations, and follow-up visits. Stratification and statistical analyses will be conducted using SPSS to evaluate differences in efficacy and safety between the two groups. The results will contribute to identifying a suitable treatment option for managing menorrhagia in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 to 39 years
2. Patients with menorrhagia
3. Incidence of breakthrough bleeding while on treatment
4. Patient with heaviness of the bleeding

Exclusion Criteria:

1. Patients with hemoglobin less than 7gm/dl
2. Patient with pelvic pathologies like uterine fibroids, suspected adenomyosis, malignancies of uterus/cervix/ovary/vagina/endometrial hyperplasia with atypia.
3. Patient with medical diseases like liver dysfunction, heart disease, migraine, stroke, renal disease, hypo/hyperthyroidism, platelet disorders or coagulopathy.
4. Patient with previous history of thrombosis; pregnancy, abortion, use of IUCDs or oral contraceptives; lactating women in first 6 months of post-natal period and hypersensitivity to the drug

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in Menstrual Blood Loss | At the end of the third treatment cycle (each cycle is 28 days).
  Menstrual blood loss will be measured using the Pictorial Blood Loss Assessment Chart (PBAC). Participants will record the number and type of sanitary products used (e.g., pads or tampons) and the degree of saturation, along with any clots passed. PBAC scores above 100 are indicative of heavy menstrual bleeding. A reduction in PBAC scores after the third treatment cycle (each cycle lasting 28 days) will be used to determine the effectiveness of the intervention.

SECONDARY OUTCOMES:
Improvement in Hemoglobin Levels | At the end of the third treatment cycle (each cycle is 28 days).
  Hemoglobin levels will be measured through venous blood samples using standard laboratory methods. Baseline levels will be recorded prior to treatment, and follow-up levels will be assessed at the end of the third treatment cycle (each cycle lasting 28 days). An increase in hemoglobin levels will indicate improved iron status and reduced anemia severity.

IPD SHARING:
Plan to Share IPD: Undecided